CLINICAL TRIAL: NCT01966718
Title: Repository Corticotropin Injection As Adjunctive Therapy In Patients With Rheumatoid Arthritis Who Have Failed At Least Three Biologic Therapies With Different Modes Of Action
Brief Title: Repository Corticotropin Injection To Treat Rheumatoid Arthritis Patients Who Have Failed Three Biologic Therapies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arthritis Treatment Center, Maryland (Other)
Responsible Party: Principal Investigator, Nathan Wei, MD, FACP, FACR:, Nathan Wei, MD, FACP, FACR, Arthritis Treatment Center, Maryland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATC 005
Record Dates: First submitted 2013-10-14; First posted 2013-10-22 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Joint pain; Repository corticotropin injection
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Repository corticotropin injection (Experimental): Repository corticotropin injection, 80 United States Pharmacopeia (USP) Units per mL, dosed as 1 mL (80 Units) subcutaneous injection every 72 hours for 12 weeks
  Interventions: Drug: Repository corticotropin injection

INTERVENTIONS:
Drug: Repository corticotropin injection — An adrenocorticotropic hormone (ACTH) analogue that stimulates the adrenal cortex to secrete cortisol, corticosterone, aldosterone, and a number of weakly androgenic substances
  Other Names: H. P. Acthar Gel

SUMMARY:
It is hypothesized that repository corticotropin injection in combination with other biologic agents will be able to provide relief of both rheumatoid arthritis and acute exacerbations of rheumatoid arthritis for patients with disease that had inadequately responded to biologics previously.

DETAILED DESCRIPTION:
Although there are many types of treatment for rheumatoid arthritis (RA) currently available, some patients have disease that is refractory to treatment and cannot achieve remission. The objective of this study is to assess the efficacy and safety of subcutaneous injections of repository corticotropin as an adjunct therapy in patients with active RA who have had an inadequate response to at least two biologic agents as well as a third agent they are currently receiving.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis of at least 2 years duration
* On at least third biologic with a different mechanism of action for at least 12 weeks
* Active disease as defined by at least 6 tender and 6 swollen joints
* Erythrocyte sedimentation rate (ESR) at least 28 mm/hr or C-reactive protein (CRP) at least 1.2 times the upper limit of normal
* Stable dose of disease modifying anti-rheumatic drug (DMARD) and prednisone for at least 4 weeks

Exclusion Criteria:

* Prior treatment with Acthar Gel
* History of intolerance or allergy to glucocorticoids
* Unstable diabetes
* Active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Wei, MD, Principal Investigator — Nathan Wei, MD dba Arthritis Treatment Center, Frederick, MD 21702 USA
Locations (1):
- Arthritis Treatment Center, Frederick, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repository Corticotropin Injection
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Rheumatoid arthritis patients who have failed at least three biologics with different methods of action
Arm/Group | Repository Corticotropin Injection
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Ritchey-Camp Articular Index
Description: Change in the Number of Joints that had Tenderness and/or Swelling According to the Ritchey-Camp Articular Index. Change was calculated using baseline and week 16 time points.
Time Frame: From baseline to week 16
Measure: Mean (Full Range); unit: joints
Units Other Than Participants: joints
Groups:
- Swollen Joints: Change in number of swollen joints participants exhibited at week 16 (Calculated by subtracting week 16 total from baseline total. Positive numbers indicate number at week 16 was less than at baseline).
- Tender Joints: Change in number of tender joints exhibited at week 16, calculated by subtracting week 16 total from baseline total.
Arm/Group | Swollen Joints | Tender Joints
Number analyzed (Participants) | 8 | 8
Number analyzed (joints) | 68 | 68
joints | 10.25 [-1 to 35] | 9 [-17 to 31]

2. Primary Outcome: Change From Baseline in the 20-item Health Assessment Questionnaire Score
Description: Subjects completed the Health Assessment Questionnaire, a 20-item scale that measures health-related quality of life. Participants are asked to rate activities on a scale from "able to do with no difficulties" to "unable to do". A score of 0 indicates the participant has no problems performing daily activities, while a score of 3 indicates that the participant is completely disabled. Scores were calculated by subtracting score at week 16 from baseline score. A positive number indicates the score went down from baseline to week 16.
Time Frame: From baseline to week 16
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Repository Corticotropin Injection
Number analyzed (Participants) | 8
units on a scale | 0.03 [-0.5 to 0.25]

3. Secondary Outcome: Change From Baseline in the Erythrocyte Sedimentation Rate (ESR)
Description: ESR was measured at baseline at week 16. Change was measured by subtracting week 16 score from baseline score. A positive number indicates that the ESR decreased
Time Frame: From baseline to week 16
Measure: Mean (Full Range); unit: mm/hr
Arm/Group | Repository Corticotropin Injection
Number analyzed (Participants) | 8
mm/hr | 1.9 [-4 to 19]

4. Secondary Outcome: Change From Baseline in the C-Reactive Protein (CRP) Level
Description: CRP was measured at Baseline and Week 16. Change was calculated by subtracting week 16 value from baseline value, with a positive value indicating a decrease from baseline.
Time Frame: From baseline to week 16
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Repository Corticotropin Injection
Number analyzed (Participants) | 8
mg/dL | 0.19 [-0.3 to 0.9]

ADVERSE EVENTS:
Time Frame: Collected at each visit (two to six week intervals) up to week 16
Arm/Group | Repository Corticotropin Injection
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repository Corticotropin Injection (N=8)
Pulmonary embolism (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repository Corticotropin Injection (N=8)
Reaction at injection site (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Development of allergies (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size (8 patients); Open label, Sampling bias cannot be excluded;Single group study; no standardization of concomitant therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No